CLINICAL TRIAL: NCT06787248
Title: Self-regulation of the mPFC Using Rt-fMRI NF Training to Enhance Positive Anticipation for Future Events
Brief Title: Real-time Neurofeedback Training of the Medial Prefrontal Cortex Based on Positive Episodic Future Thinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BAM_lab_NF_05
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Neurofeedback
Keywords: real-time neurofeedback; episodic future thinking; mPFC

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback training (Experimental): Subjects in the neurofeedback training group are instructed to regulate their medial prefrontal cortex activity based on the visual neurofeedback.
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure
- Control (Sham Comparator): Subjects in the sham control group receive the same instruction but perform the regulation based on neurofeedback from an unrelated region (i.e. primary motor cortex) which is not involved in episodic future thinking (a controlled sham region).
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure

INTERVENTIONS:
Procedure: real-time fMRI sham-controlled neurofeedback training procedure — real-time fMRI neurofeedback training procedure running on the Turbo Brain voyager (TBV) 4.2 software (Brain Innovation, Maastricht, The Netherlands)

SUMMARY:
Randomized active-sham controlled between-subject real-time fMRI neurofeedback trial aiming to modulate activity in the medial prefrontal cortex (mPFC) to improve subjective positive anticipation.

DETAILED DESCRIPTION:
A randomized double-blind sham-controlled between-subject design using real-time fMRI neurofeedback. In a randomized order, a total of 60 healthy subjects will be recruited and assigned (1) experimental group (EG; N=30), which receives real neurofeedback from the left medial prefrontal cortex (mPFC), or (2) control group (CG; N=30) which receives sham neurofeedback from the primary motor cortex (M1). Neurofeedback training consists of 1 baseline session without feedback, 4 training sessions with real-time feedback, and and 1 transfer session without feedback. Resting state fMRI will be employed to explore neural effects. Objectives are to determine (1) if subjects in the neurofeedback (NF) group can gain volitional control over the mPFC activation using positive episodic regulation strategy, (2) whether successful increased modulation of the mPFC could enhance positive anticipation for future events and motivation (using the Effort-Expenditure for Reward Task, EEfRT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Psychiatric or Neurological Disorder
* Contraindications for MRI
* Regular use of psychotropic substances (medication, drugs)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Neural activity of the medial prefrontal cortex (mPFC) based on blood oxygen level-dependent (BOLD) signal | 1 hour
  Training-induced changes in mPFC activity will be assessed by analyzing BOLD-level activation of the mPFC

SECONDARY OUTCOMES:
Training-related changes in anticipated pleasure | 1 hour
  Participants will be required to rate the anticipated pleasantness of future events using a Likert Scale ranging from 1 to 9 (1 = not at all pleasant) and 9 = very pleasant).
Training-related changes in motivational effort | 1 hour
  Training-induced changes in motivational effort as measured by the Effort Expenditure for Rewards Task (EEfRT)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Corresponding individual level data will be made available upon request